CLINICAL TRIAL: NCT04272905
Title: Recording by Patients and Relatives/Friends in the Maternity Unit - Patient and Staff Knowledge/Attitudes
Brief Title: Recording by Patients and Relatives/Friends in the Maternity Unit
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W 19/016; 258908 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2020-02-06; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Knowledge, Attitudes, Practice; Maternity; Health Personnel Attitude; Healthy
Keywords: Knowledge; Attitudes; Recording; Maternity
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maternity patients: * > 18 years
  * Post-natal following any form of delivery
  * Between 4 and 48 hours after delivery
  * Able to understand English adequately to give consent and complete the questionnaire
  Interventions: Other: Non-interventional study
- Maternity Unit Staff: * Doctors, midwives and other staff
  * Work on labour ward
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — The participants will be asked to complete a questionnaire on their knowledge of, and attitudes towards the recording of patient care by patients or relatives/friends in the maternity unit. An investigator will be immediately available to facilitate completion of the survey and assist with understanding of the questions. The data recorded will be a mixture of nominal data (selections from a number of options using a tickbox) or ordinal (as above, but graded e.g. yes / yes with qualifiers / no). Free text will be coded and presented as nominal data or presented verbatim to illustrate points that arise.

SUMMARY:
Increasingly, patients are keen to record aspects of their medical care, especially in obstetrics and paediatrics. The knowledge of patients and staff in relation to this area is thought to be variable. In addition, the attitudes of patients and staff regarding this practice has not been well studied. This study aims to gather information on patients' use of recording devices to capture audio recordings, photographs or videos. Furthermore it aims to assess patient and staff knowledge and attitudes in relation to this area.

This study will involve patients who have recently delivered a baby on the maternity unit or obstetric theatre completing a questionnaire. They will be approached by a study investigator and the study explained. They will then complete a consent form if they are happy to proceed. Following this they will complete the questionnaire.

It will also involve the surveying of staff, who will be approached by a study investigator when not directly involved in the clinical care of patients. They will also complete a consent form if they are happy to proceed and then complete the questionnaire.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the knowledge and attitudes of both patients and staff towards the recording by patients/relatives/friends within the obstetric environment.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Post natal following any form of delivery
* Between 4 and 48 hours after delivery
* Able to understand English adequately to give consent and complete the questionnaire

Exclusion Criteria:

- Women experiencing complications affecting themselves or their babies will be excluded if it is felt that approaching them for potential recruitment might be overly intrusive.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As above.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Knowledge and attitudes of both patients and staff towards the recording by patients/relatives/friends within the maternity unit and obstetric theatre environment. | Cross-sectional design: Participants are expected to be in the study for 15 minutes approx.
  Staff and patients will be asked to complete an unvalidated questionnaire titled "Recording by patients and relatives/friends in the maternity unit", which is expected to take 10-15 minutes to complete. Please note that one questionnaire has been adapted for patients and another one for staff. Both contain 4 sections. The sections in the patients' questionnaire are: Background, Your experience of recording, Guidelines on recording and Your opinions regarding recording. The sections in the staff's questionnaire are: Background, Your experience of recording, Knowledge and Attitudes.
  Data will be presented using descriptive statistics: Number (%) ± 95% CI for nominal data and median (IQR [range]) for ordinal data as appropriate.

SECONDARY OUTCOMES:
Group differences between the knowledge and attitudes of patients and staff regarding what is acceptable to record and appropriate uses of recordings. | Data analysis will be completed and reported within an average of one year.
  Analytic statistics will be performed to compare differences in the results of the unvalidated questionnaire between the two groups (patients and staff) using the chi-squared/Fisher's exact test for nominal data and Mann-Whitney U-test for ordinal data, taking p < 0.05 to denote statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula McHugh, MB BCh BaO, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsulukidze M, Durand MA, Barr PJ, Mead T, Elwyn G. Providing recording of clinical consultation to patients - a highly valued but underutilized intervention: a scoping review. Patient Educ Couns. 2014 Jun;95(3):297-304. doi: 10.1016/j.pec.2014.02.007. Epub 2014 Mar 3. PMID 24630697
- [Background] NHS Protect. Patients recording NHS staff in health and social care settings. 2016.
- [Background] Care Quality Commission. Thinking about using a hidden camera or other equipment to monitor someone's care. 2015.
- See also: Recording video has never been so easy or effortless — https://www.pocket-lint.com/phones/news/131351-10-tips-for-recording-better-video-with-your-smartphone
- See also: The Care Quality Commission discusses using cameras or other recording equipment to check somebody's care — https://www.cqc.org.uk/sites/default/files/20150212_public_surveillance_leaflet_final.pdf
- See also: Digital dilemmas - Patients recording consultations — http://www.medicalprotection.org/uk/articles/digital-dilemmas-patients-recording-consultations
- See also: Photographers Rights And The Law In The UK - The law and photography. — http://www.urban75.org